CLINICAL TRIAL: NCT04928027
Title: Self-Reports of Executive Functions in Persons With Parkinson's Disease and Their Significant Others
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Old Dominion University (Other)
Responsible Party: Principal Investigator, Jane Roitsch, Assistant Professor, Old Dominion University
Other Study IDs: EFs and PD
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Parkinsonism or Parkinson's Disease Nos
MeSH Terms: conditions — Parkinsonian Disorders; Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons with PD: Adults with PD will be provided with email link to complete the Comprehensive Executive Function Inventory-Self-Assessment
- Significant Others of those with PD: Adults whose significant other has a diagnosis of PD will be provided with email link to complete the Comprehensive Executive Function Inventory-Observer report

SUMMARY:
The investigators are conducting a study to compare the self-reports of executive functions (that is to say, what role cognitive processes such as working memory and attention) in persons with Parkinson's Disease to the reports of executive functions completed by their significant others.

To conduct this study, the investigators need the participation of persons who are diagnosed with Parkinson's Disease and their significant others.

DETAILED DESCRIPTION:
The purpose of this study is to explore the relationship between the self-reported executive functions (EFs) in persons with Parkinsons disease (PD) and their significant others. Executive functions include basic cognitive processes such as attention, inhibition, working memory, and cognitive flexibility. As this proposed study will test not only cognitive functioning, but specific aspects of it (i.e., EFs) without excluding persons with PD who have identified cognitive impairments, outcomes gathered could provide valuable information to better assist all types of persons with PD. Comparing their self-reported EFs to the EF ratings completedy by their signifiant others can help determine if a disparity exists between self-perceptions and actual observed EF abilties. This study would assess EFs through inhibition responses of participants via computerized versions the Comprehensive Executive Function Inventory-Adult Self-Report and Observer forms.

ELIGIBILITY:
Inclusion Criteria:

* For persons with PD,confirmed diagnosis of PD) For significant others - relationship with person with PD

Exclusion Criteria:All participants will be screened to ensure they do not have:

* any known cognitive disorders other than those associated with PD
* impairments in vision that would affect their ability to safely participate in the study
* recent history of neuromuscular injury/ damage that could affect their ability to complete the CEFI
* the participant will be excluded if he or she is unable to follow commands well enough to complete the CEFI

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's group: Adults with a Parkinson's disease diagnosis and their significant others.
  Healthy elderly: no history of neurologic disease (e.g., stroke, traumatic brain injury)
  Both groups:
  Age 30-79 years with no history of other neurologic diseases, orthopedic, or arthritic conditions that preclude ability to walk
  Some of the earliest cognitive symptoms of Parkinsonism involve executive function deficits (e.g., working memory, cognitive flexibility, planning; Williams-Gray, Foltynie, Lewis, and Barker, 2006). What is less understood, however, is whether a relationship exists between the self-reported EFs in persons with Parkinsonism and their significant others. The need for research to investigate the relationship between EFs in persons with Parkinsonism is evident in the limited body of literature currently available.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-06-08 (Estimated); Study Completion 2022-06-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of EF outcomes | 1 year
  Results of the self-reports of persons with PD and their Significant Others will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No other researchers will received participant data information